CLINICAL TRIAL: NCT01980992
Title: Oral Immunotherapy for Wheat Allergy
Acronym: Wheat OIT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hugh A Sampson, MD (Other)
Responsible Party: Sponsor-Investigator, Hugh A Sampson, MD, Dean for Translational Biomedical Sciences, Director, Jaffe Food Allergy Institute, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 11-0197; FAI001 (Other: Jaffe Food Allergy Institute)
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Wheat Allergy
Keywords: Food Allergy; Wheat Allergy; Oral Immunotherapy
MeSH Terms: conditions — Wheat Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wheat OIT (Active Comparator): Active treatment participants receive Vital Wheat Gluten, and have up to four oral food challenges as directed by the protocol.
  Interventions: Drug: Wheat OIT
- Placebo (Placebo Comparator): Placebo for Vital Wheat Gluten followed by crossover to open-label active therapy (Vital Wheat Gluten), and up to three oral food challenges as directed by the protocol.
  Interventions: Drug: Wheat OIT

INTERVENTIONS:
Drug: Wheat OIT — Vital Wheat Gluten dispensed by the central manufacturer. Study product will be dispensed in vials for low doses, capsules for mid-range doses, and bulk powder with dosing scoops for the higher doses.
  Other Names: Vital Wheat Gluten

SUMMARY:
This study is being done to learn about the medical effects, the safety, and the immunologic effects of Wheat Oral Immunotherapy (OIT) treatment. The goal of the study is to find out whether subjects can develop the ability to eat wheat (the food allergen) regularly without allergic symptoms after stopping the study treatment.

DETAILED DESCRIPTION:
Food allergy affects 6-8 percent of children in the United States. Wheat is one of the eight most common foods inducing allergic reactions in the US. Current treatment for food allergy is complete avoidance of the food and to carry antihistamines and self-injectable epinephrine if an accidental reaction occurs. However, accidental exposure to allergens in processed foods may be difficult to avoid. Currently, several therapeutic strategies are being investigated to prevent and treat food allergies. Since immunotherapy injections for food allergy are associated with a high rate of allergic reactions, alternate approaches to treatment are needed. Oral (by mouth) immunotherapy (OIT) is one approach that has been tried in some studies in the treatment of food allergies. The intent of the study is to examine the clinical effects and safety of wheat OIT. This study will last 2 years. All eligible subjects will receive a wheat oral food challenge (OFC). Those who react to 1923mg or less of vital wheat gluten will be randomized to Wheat OIT or a placebo. All eligible and enrolled subjects will have a 1-year and 2-year OFC. Placebo subjects will crossover to Wheat OIT at the 1-year time point. At selected visits, blood and urine collection, physical examination, prick skin tests, and atopic dermatitis and asthma evaluations will occur.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-30 years either sex, any race, any ethnicity
* Positive Prick Skin Test to wheat greater than 3mm compared to control and/or a wheat specific IgE >= 0.35 kUA/L
* Positive baseline challenge to wheat (<= 1923 mg of vital wheat gluten)
* Written informed consent from subject and/or parent/guardian
* Written assent from all subjects as appropriate
* All females of child bearing age must be using appropriate birth control

Exclusion Criteria:

* History of anaphylaxis to wheat resulting in hypotension, neurological compromise or mechanical ventilation
* Known allergy to corn
* Known celiac disease
* Chronic disease (other than asthma, atopic dermatitis, rhinitis) requiring therapy (e.g., heart disease, diabetes)
* Active eosinophilic gastrointestinal disease in the past two years
* Participation in any interventional study for the treatment of food allergy in the past 6 months
* Subject is on "build-up phase" of immunotherapy (i.e., has not reached maintenance dosing). Subjects tolerating maintenance allergen immunotherapy can be enrolled.
* Severe asthma, uncontrolled mild or moderate asthma. More information on this criterion can be found in the protocol.
* A burst of oral, IM or IV steroids of more than 2 days for an indication other than asthma in the past 1 month
* Inability to discontinue antihistamines for initial day escalation, skin testing or OFC
* Use of omalizumab or other non-traditional forms of allergen immunotherapy or immunomodulator therapy (not including corticosteroids) or biologic therapy within the past year
* Use of beta-blockers (oral), angiotensin-converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARB) or calcium channel blockers
* Use of investigational drug within 90 days or plan to use investigational drug during the study period
* Pregnancy or lactation

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2013-10; Primary Completion 2015-11 (Actual); Study Completion 2017-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh A Sampson, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Hugh A Sampson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - Stanford University School of Medicine, Stanford, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began November 2013 and was completed in November 2014
Groups:
- Placebo Then High Dose Group: 52 weeks placebo, then crossed over to active wheat oral immunotherapy (OIT) to a maximum dose of 3870mg wheat powder (2748 mg wheat protein). Placebo subjects who were crossed over received a higher maintenance dose than the Wheat OIT subjects. After this group received 52 weeks of active wheat OIT treatment, they then completed a Week 52 7443mg wheat protein oral food challenge (OFC).
- Wheat OIT: 2 years on active wheat oral immunotherapy (OIT) with maximum maintenance dose 2035mg wheat powder (1445mg wheat protein), then completed Year 2 7443 mg wheat protein desensitization oral food challenge (OFC); those that passed this OFC stopped active OIT treatment for 8-10 weeks and then completed the Year 2 7443 mg wheat protein tolerance OFC.
Period: 52 Weeks Blinded Study Treatment
Arm/Group | Placebo Then High Dose Group | Wheat OIT
Started | 23 | 23
Completed | 21 | 19
Not Completed | 2 | 4
Not completed — Dosing Symptoms | 0 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Non-compliance | 1 | 0
Period: 52 Weeks Open Label Active Wheat OIT
Arm/Group | Placebo Then High Dose Group | Wheat OIT
Started | 21 | 19
Completed | 18 | 18
Not Completed | 3 | 1
Not completed — Dosing Symptoms | 2 | 0
Not completed — Non-compliance | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then High Dose Group | Wheat OIT | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Median (Full Range); unit: years] | 8.7 [4.2 to 22.3] | 8.6 [4.6 to 18.4] | 8.7 [4.2 to 22.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 18 | 18 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 23 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 15 | 29
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Wheat IgE [Median (Inter-Quartile Range); unit: kUA/L] — Amount of serum wheat-specific immunoglobulin E (IgE). Individuals with a wheat IgE of <0.35 kUA/L are considered not to be sensitized to wheat. The limits of detection for the wheat IgE assay were 0.1 to 100 kUA/L. Values below the limit of detection were set to 0.05 kUA/L and those above the limit of detection were set to 101 kUA/L.
  kUA/L | 86.8 [63.7 to 101.0] | 94.1 [45.0 to 101.0] | 88.4 [51.9 to 101.0]
Wheat IgG4 [Median (Inter-Quartile Range); unit: mgA/L] — Amount of immunoglobulin G4 (IgG4). The limits of detection for the wheat IgG4 assay were 0.1 to 30 mgA/L. Values below the limit of detection were set to 0.05 mgA/L and those above the limit of detection were set to 31 mgA/L for wheat IgG4.
  mgA/L | 4.6 [2.5 to 8.6] | 2.9 [1.7 to 10.2] | 4.2 [2.1 to 9.9]
Wheat Skin Prick Test [Mean (Standard Deviation); unit: mm] — This score is calculated by subtracting the size of the saline wheal (in mm) from the size of the wheat wheal (in mm) observed for a skin prick test. Individuals with a wheat skin prick test score of < 3 mm are considered to have a negative result.
  mm | 6.8 (2.8) | 5.3 (3.4) | 6.1 (3.2)
Wheat OFC Dose at First Symptom [Median (Inter-Quartile Range); unit: mg protein] | 13.0 [3.0 to 43.0] | 43.0 [13.0 to 443.0] | 13.0 [3.0 to 143.0]
Wheat OFC Successfully Consumed Dose [Median (Inter-Quartile Range); unit: mg protein] | 43.0 [3.0 to 143.0] | 43.0 [13.0 to 143.0] | 43.0 [3.0 to 143.0]
Maximum Initial Escalation Day Dose [Median (Full Range); unit: mg powder] | 12.0 [3.0 to 12.0] | 12.0 [6.0 to 12.0] | 12.0 [3.0 to 12.0]

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Desensitized Participants as Measured by the Ability to Consume at Least 4443 mg of Wheat Protein During a 7443 mg Wheat Protein Oral Food Challenge (OFC) Performed 1 Year After Initiating Treatment.
Description: Determine in wheat allergic children, whether relative to placebo, daily oral administration of Vital Wheat Gluten escalated to a maximum of 2035 mg/day of Vital Wheat Gluten increases desensitization as measured by consuming without dose limiting symptoms 4443 mg of wheat protein on a 7443 mg wheat protein OFC performed 1 year after initiating treatment.
Time Frame: 1 Year
Population: All randomized participants were included.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: 52 weeks placebo, then crossed over to active wheat oral immunotherapy (OIT) to a maximum dose of 3870mg wheat powder (2748 mg wheat protein). Placebo subjects who were crossed over received a higher maintenance dose than the Wheat OIT subjects. After this group received 52 weeks of active wheat OIT treatment, they then completed a week 52 7443mg wheat protein oral food challenge (OFC).
Arm/Group | Placebo | Wheat OIT
Number analyzed (Participants) | 23 | 23
Participants | 0 | 12

2. Secondary Outcome: Number of Subjects Who Successfully Consume a Wheat Protein Oral Food Challenge
Description: The number of subjects who successfully consume a 7443 mg wheat protein oral food challenge (OFC) 8-10 weeks after therapy discontinuation and after passing the 7443 mg wheat protein OFC at the 2 year time point.This OFC will only be administered to subjects in the initial active treatment group.
Time Frame: 8 to 10 weeks after passing the 2 Year OFC
Population: This is not applicable for the Placebo Crossover subjects as they did not complete at 2 Year Tolerance OFC per the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Then High Dose Group | Wheat OIT
Number analyzed (Participants) | 0 | 23
Participants | 0 | 3

3. Secondary Outcome: Number of Subjects Who Achieve the Targeted Maintenance Dose of Wheat OIT
Description: The number of subjects who achieve the targeted maintenance dose of wheat OIT during the desensitization phase of the study. For Wheat OIT group, reached target dose of 2035 mg wheat powder/1445 mg wheat protein. For placebo group, reached target dose of 2035 mg placebo powder.
Time Frame: 44 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Then High Dose Group | Wheat OIT
Number analyzed (Participants) | 23 | 23
Participants | 21 | 19

4. Secondary Outcome: Number of Subjects That Achieve Desensitization in the Placebo Cross Over Group
Description: The number of subjects that achieve desensitization in the placebo cross over group after 1 year of dosing. Able to consume at least 4443 mg wheat protein on the Week 52 Crossover OFC (4443 mg wheat protein is the amount that was used for the primary endpoint).
Time Frame: 2 Years
Population: Two Placebo subjects did not crossover. This outcome measure is only for the Placebo crossover group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Then High Dose Group
Number analyzed (Participants) | 21
Participants | 14

5. Secondary Outcome: Incidence of All Serious Adverse Events During the Study.
Time Frame: 1 year and 2 Years
Population: Data was available for 22 participants in the Wheat OIT group and 21 participants for the Placebo Crossover group at the end of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Wheat OIT Before 1 Year: During the first year of 2 years on active wheat oral immunotherapy (OIT) with maximum maintenance dose 2035mg wheat powder (1445mg wheat protein), then completed Year 2 7443 mg wheat protein desensitization oral food challenge (OFC); those that passed this OFC stopped active OIT treatment for 8-10 weeks and then completed the Year 2 7443 mg wheat protein tolerance OFC.
- Placebo Before 1 Year: During the first year of 52 weeks placebo, then crossed over to active wheat oral immunotherapy (OIT) to a maximum dose of 3870mg wheat powder (2748 mg wheat protein). Placebo subjects who were crossed over received a higher maintenance dose than the Wheat OIT subjects. After this group received 52 weeks of active wheat OIT treatment, they then completed a Week 52 7443mg wheat protein oral food challenge (OFC).
- Wheat OIT After 1 Year: 2 years on active wheat oral immunotherapy (OIT) with maximum maintenance dose 2035mg wheat powder (1445mg wheat protein), then completed Year 2 7443 mg wheat protein desensitization oral food challenge (OFC); those that passed this OFC stopped active OIT treatment for 8-10 weeks and then completed the Year 2 7443 mg wheat protein tolerance OFC.
- Placebo Crossover: 52 weeks placebo, then crossed over to active wheat oral immunotherapy (OIT) to a maximum dose of 3870mg wheat powder (2748 mg wheat protein). Placebo subjects who were crossed over received a higher maintenance dose than the Wheat OIT subjects. After this group received 52 weeks of active wheat OIT treatment, they then completed a Week 52 7443mg wheat protein oral food challenge (OFC).
Arm/Group | Wheat OIT Before 1 Year | Placebo Before 1 Year | Wheat OIT After 1 Year | Placebo Crossover
Number analyzed (Participants) | 23 | 23 | 22 | 21
Participants | 0 | 3 | 1 | 1

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Wheat OIT Before 1 Year; Wheat OIT After 1 Year: 2 years on active wheat oral immunotherapy (OIT) with maximum maintenance dose 2035mg wheat powder (1445mg wheat protein), then completed Year 2 7443 mg wheat protein desensitization oral food challenge (OFC); those that passed this OFC stopped active OIT treatment for 8-10 weeks and then completed the Year 2 7443 mg wheat protein tolerance OFC.
- Placebo Before 1 Year; Placebo Crossover: 52 weeks placebo, then crossed over to active wheat oral immunotherapy (OIT) to a maximum dose of 3870mg wheat powder (2748 mg wheat protein). Placebo subjects who were crossed over received a higher maintenance dose than the Wheat OIT subjects. After this group received 52 weeks of active wheat OIT treatment, they then completed a Week 52 7443mg wheat protein oral food challenge (OFC).
Arm/Group | Wheat OIT Before 1 Year | Placebo Before 1 Year | Wheat OIT After 1 Year | Placebo Crossover
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 3/23 | 1/22 | 1/21
Other Adverse Events (participants affected / at risk) | 23/23 | 21/23 | 18/22 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wheat OIT Before 1 Year (N=23) | Placebo Before 1 Year (N=23) | Wheat OIT After 1 Year (N=22) | Placebo Crossover (N=21)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wheat OIT Before 1 Year (N=23) | Placebo Before 1 Year (N=23) | Wheat OIT After 1 Year (N=22) | Placebo Crossover (N=21)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 10 (48) | 3 (27) | 2 (22) | 7 (79)
Urticaria (Skin and subcutaneous tissue disorders) | 11 (57) | 9 (16) | 3 (13) | 12 (49)
Flatulence (Gastrointestinal disorders) | 1 (4) | 1 (16) | 1 (8) | 0 (0)
Nausea (General disorders) | 2 (3) | 1 (2) | 2 (6) | 0 (0)
Vomiting (General disorders) | 8 (25) | 0 (0) | 1 (5) | 7 (20)
Gastroenteritis (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Rhinitis allergic (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (8) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Abdominal discomfort (Gastrointestinal disorders) | 16 (484) | 6 (28) | 6 (74) | 13 (146)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (20) | 2 (6) | 1 (5) | 2 (11)
Dyspepsia (Gastrointestinal disorders) | 1 (8) | 0 (0) | 1 (1) | 3 (3)
Gastrontestinal disorder (Gastrointestinal disorders) | 17 (172) | 11 (57) | 5 (14) | 16 (153)
Gastrooescophageal refluz disease (Gastrointestinal disorders) | 2 (8) | 1 (1) | 0 (0) | 1 (5)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Oral mucosal eruption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Saliva altered (Gastrointestinal disorders) | 1 (17) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 4 (5) | 2 (2) | 2 (2)
Chest discomfort (General disorders) | 4 (85) | 3 (3) | 1 (1) | 4 (13)
Chest pain (General disorders) | 1 (5) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 4 (5) | 1 (1) | 3 (4) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 2 (2) | 3 (4) | 1 (1)
Hypersensitivity (Immune system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Croup infectious (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 2 (3)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 5 (11) | 7 (10) | 4 (4) | 10 (17)
Viral infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3) | 1 (1) | 3 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 3 (3) | 0 (0) | 0 (0)
nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (7) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (55) | 5 (12) | 4 (7) | 8 (32)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (10) | 0 (0) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 (126) | 2 (2) | 2 (12) | 6 (31)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (304) | 7 (10) | 6 (27) | 17 (200)
Rhimorrhoea (Respiratory, thoracic and mediastinal disorders) | 16 (157) | 8 (16) | 4 (14) | 11 (45)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 5 (9) | 0 (0) | 5 (10)
dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (121) | 13 (311) | 1 (8) | 13 (347)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 1 (1) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1) | 0 (0) | 2 (2)
Flashing (Vascular disorders) | 6 (40) | 7 (9) | 1 (2) | 10 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes